CLINICAL TRIAL: NCT02955758
Title: A Phase 2 Trial of Pembrolizumab in Metastatic Non-squamous NSCLC Examining Circulating Tumor DNA Levels as a Surrogate Biomarker of Response
Brief Title: Pembrolizumab in Patients With Metastatic Non-squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joel Neal (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Joel Neal, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-37785; NCI-2016-01311 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-37785 (Other: Stanford IRB); LUN0085 (Other: OnCore)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Non-Squamous Non-Small Cell Lung Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV, 200mg fixed dose, every 3 weeks
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with non-squamous non-small cell lung cancer which has spread to other places in the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate circulating tumor DNA (ctDNA) levels measured using cancer personalized profiling by deep sequencing (CAPP-Seq) with radiographic tumor assessments using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria in patients with metastatic non-squamous non-small cell lung cancer (NSCLC) treated with pembrolizumab.

SECONDARY OBJECTIVES:

I. To correlate PD-L1 assessment on pre-treatment tumor samples with objective response using RECIST v1.1 criteria in patients with metastatic non-squamous NSCLC treated with pembrolizumab.

II. To determine the overall response rate (ORR) using RECIST v1.1 criteria in patients with metastatic non-squamous NSCLC treated with pembrolizumab.

III. To determine the progression-free survival (PFS) using RECIST v1.1 in patients with metastatic non-squamous NSCLC treated with pembrolizumab.

IV. To determine the overall survival (OS) in patients with metastatic non-squamous NSCLC treated with pembrolizumab.

V. To determine the safety and tolerability of pembrolizumab in patients with metastatic non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Has a pathologically proven recurrent or metastatic non squamous non small cell lung cancer
2. (a) Previously received at least one line of prior systemic therapy for metastatic disease.

   i. If the patient has a sensitizing EGFR mutation or ALK rearrangement, the patient must have received at least one prior targeted therapy for metastatic disease (ie, EGFR TKI therapy or ALK TKI therapy, respectively).

   ii. There is no limit on prior therapies allowed. Patients must have completed previous treatment (including other investigational therapy) in greater than or equal to the following times prior to initiation of trial treatment:
   1. Anti cancer monoclonal antibody (mAb) therapy must be completed ≥ 3 weeks prior to trial treatment
   2. Chemotherapy administered in a daily or weekly schedule must be completed ≥ 1 week prior to trial treatment
   3. Chemotherapy administered in an every 2 week schedule must be completed ≥ 2 weeks prior to trial treatment
   4. Chemotherapy administered in an every 3 week schedule must be completed ≥ 3 weeks prior to trial treatment
   5. Targeted small molecule therapy must be completed ≥ 1 week prior to trial treatment OR (b) Have not received prior systemic therapy for their cancer in recurrent or metastatic setting, AND have a tumor with Tumor Proportion Score (TPS) ≥ 50% as measured by 22C3 PD L1 IHC test, AND no evidence of a sensitizing EGFR mutation or ALK rearrangement.
3. Prior radiation therapy allowed as long as completed in the following times prior to initiation of trial treatment:

   1. Definitive curative intent radiation ≥ 3 weeks prior to trial treatment
   2. Palliative body radiation ≥ 1 week prior to trial treatment
   3. Stereotactic brain radiation ≥ 1 week prior to trial treatment
   4. Whole brain radiation ≥ 2 weeks prior to trial treatment
4. Patients with previously treated (with radiation or surgery) brain metastases that are stable are allowed. Patients with stable or progressing metastases must have metastases ≤ 1.5 cm, be asymptomatic, and either not be on steroids or be on 10 mg prednisone equivalent or less.
5. Has measurable disease based on RECIST v1.1 criteria
6. Is medically able and willing to undergo needle biopsy of a tumor lesion. PD L1 expression is not required to enroll in the trial.
7. Has life expectancy ≥ 3 months
8. Ability to understand and the willingness to sign a written informed consent document.
9. ≥ 18 years of age on day of signing informed consent
10. ECOG performance status of 0 or 1 (Appendix A)
11. Adequate organ function:

    1. Absolute neutrophil count (ANC) ≥ 1,000/mcL
    2. Platelets ≥ 75,000/mcL
    3. Hemoglobin ≥ 8 g/dL
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 50 mL/min for patient with creatinine levels > 1.5 x institutional ULN
    5. Serum total bilirubin ≤ 1.5 x ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN
    6. AST (SGOT) and ALT (SGPT) ≤ 3 x ULN OR ≤ 5 x ULN for patients with liver metastases
12. Female patients of childbearing potential must have a negative urine or serum pregnancy test prior to the first dose of trial treatment. They must also agree to two barrier methods or a barrier method plus a hormonal method, or agree to abstain from heterosexual activity, for the course of the study through 120 days after the last dose of trial treatment. Females who have been surgically sterilized or are free from menses for > 1 year (postmenopausal) may enroll.
13. Male patients with a female partner of childbearing potential should agree to use a barrier method of contraception, or agree to abstain from heterosexual activity for the course of the study through 120 days after the last dose of trial treatment.

Exclusion Criteria:

1. Is currently receiving another investigational therapy
2. Has received prior anti PD 1 or anti PD L1 therapy
3. Has clinically significant toxicities from previous anti cancer therapy that have not resolved, or have not stabilized at a new baseline
4. Has undergone a surgical procedure involving general anesthesia within 2 weeks of starting trial treatment, or has inadequate healing or recovery from complications of surgery prior to starting trial treatment. This does not apply to low risk procedures such as thoracentesis; paracentesis; chest tube/PleurX catheter placement; line placement; needle biopsy of tumor; and bronchoscopy.
5. Is receiving high dose systemic steroid therapy within 3 days of trial treatment. Topical and intraarticular steroid injections are allowed, as are physiologic doses of systemic steroids (≤ 10 mg of prednisone equivalent daily).
6. Has carcinomatous meningitis as determined by positive CSF cytology
7. Has known active additional malignancy that is undergoing active treatment.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, supra physiologic doses of systemic corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin; or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Asthma; type I diabetes mellitus; hypothyroidism; and vitiligo are allowed.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator. This includes known active tuberculosis; Grade 3 active infection; history of allogeneic bone marrow transplant or solid organ transplant; known history of Human Immunodeficiency Virus (HIV); known active Hepatitis B (eg, Hep B DNA positive in prior 3 months) or known active Hepatitis C (eg, HCV RNA [qualitative] is detected in prior 3 months).
10. Known active interstitial lung disease, or current (non infectious) pneumonitis or history of (non infectious) pneumonitis that required oral steroids.
11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neal, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Tumor-informed CAPP-Seq ctDNA Analysis With Radiologic Tumor Assessments
Description: Circulating tumor DNA (ctDNA) levels will be measured using Cancer personalized profiling by deep sequencing (CAPP Seq) with radiographic tumor assessments using RECIST v1.1 criteria in patients with metastatic NSCLC treated with pembrolizumab. ctDNA will be measured as percentage of total circulating free DNA. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Population: All patients enrolled and treated
Measure: Number; unit: Percent Accuracy
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 25
Percent Accuracy
  Complete Response (CR)/Partial Response (PR): number analyzed (Participants) | 2
  Complete Response (CR)/Partial Response (PR) | 100
  Stable Disease (SD): number analyzed (Participants) | 9
  Stable Disease (SD) | 66
  Progressive Disease (PD): number analyzed (Participants) | 7
  Progressive Disease (PD) | 100
  Non-Evaluable (NE): number analyzed (Participants) | 7
  Non-Evaluable (NE) | NA — Pre/post ctDNA and Radiographic response need to be evaluable to measure primary outcome. No evaluable somatic mutations identified in 3 patients, no evaluable post-treatment plasma available in 3 patients, and follow up radiographic response not performed in 1 patient.

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) defined as proportion of complete responses + partial responses will be measured using RECIST v1.1 criteria
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 25
participants | 2

3. Secondary Outcome: PFS Measured Using RECIST v1.1 Criteria
Description: Progression-free survival (PFS) will be measured from the time of first treatment with pembrolizumab to the time of radiographic progression, unequivocal clinical progression, or death from any cause, whichever comes earlier
Time Frame: From the time of first treatment with pembrolizumab to the time of progression or death from any cause, whichever comes earlier, assessed up to 2 years
Population: PFS Evaluable Patients by RECIST 1.1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 25
Months | 2.6 [1.3 to 4.9]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival of all treated participants
Time Frame: From the time of first treatment with pembrolizumab to the time of death, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 25
Months | 13.3 [10.3 to 27.8]

5. Secondary Outcome: Incidence of Adverse Events Graded According to Common Terminology Criteria for Adverse Events Version 4.03
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=25)
Worsening dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
Recurrence of bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
worsening of oncologic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bacterial pneumonia (Infections and infestations) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
Worsening bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Worsening pericardial effusion with Tamponade (Cardiac disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
pain (General disorders) | 1 (1)
altered mental status (Nervous system disorders) | 1 (1)
Craniotomy (Surgical and medical procedures) | 1 (1) — Right parietal craniotomy for resection of tumor
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab) (N=25)
intermittent blurry vision (Eye disorders) | 1 (2)
visual changes (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Worsening abdominal pain (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Worsening vomiting (Gastrointestinal disorders) | 1 (1)
Worsening diarrhea (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Post-operative abdominal pain (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Worsening back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Upper back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
General back pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Left sided rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left foot discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening left hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Right-sided muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Renal failure and altered mental status (Musculoskeletal and connective tissue disorders) | 1 (1)
Runny nose (allergies) (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Musculoskeletal and connective tissue disorders) | 1 (1)
Malaise (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Venous distention (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Contrast allergic reaction (Immune system disorders) | 1 (1)
Elevated AST (Investigations) | 1 (2)
Elevated creatinine (Investigations) | 1 (1)
Neutrophilia (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Worsening decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Right heel infection (Infections and infestations) | 1 (1)
Rash acneiform on shoulder (Infections and infestations) | 1 (1)
Rash acneiform on face (Infections and infestations) | 1 (1)
Rash acneiform (Infections and infestations) | 1 (1)
Rash acneiform on chest (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Rash acneiform on back (Infections and infestations) | 1 (1)
Rash acneiform on buttocks (Infections and infestations) | 1 (1)
Rash acneiform on feet (Infections and infestations) | 1 (1)
Rash acneiform on arms (Infections and infestations) | 1 (1)
Neck pain (Infections and infestations) | 2 (3)
Worsening muscle weakness (Infections and infestations) | 1 (1)
Rib pain (Infections and infestations) | 1 (2)
Left shoulder pain (Infections and infestations) | 2 (2)
Post-surgical chest pain (Infections and infestations) | 1 (1)
Intermittent RUE muscle cramps (Infections and infestations) | 1 (1)
Non-cardiac chest pain (Infections and infestations) | 1 (1)
Cramps (arms) (Infections and infestations) | 1 (1)
Cramps (legs) (Infections and infestations) | 1 (1)
Weakness in right hand (Infections and infestations) | 1 (1)
Intermittent achiness (Infections and infestations) | 1 (1)
Arthritic pain in hands (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Anterior chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Possible tuberculosis reactivation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Lower extremity edema (General disorders) | 4 (5)
Fatigue (General disorders) | 2 (6)
Neuropathy (General disorders) | 1 (1)
Worsening fatigue (General disorders) | 3 (3)
Post-biopsy pain (left rib) (General disorders) | 1 (1)
Neuropathy (Left chest wall) (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hydrocephalus (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Worsening headache (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Itchy skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hot flashes (Vascular disorders) | 1 (1)
Worsening hot flashes (Vascular disorders) | 1 (1)
Possible temporal arteritis (Vascular disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT02955758/Prot_SAP_000.pdf